CLINICAL TRIAL: NCT02012036
Title: OPTIC-III Prospective Non-Interventional Study To Optimize Photodynamic TUR-B In Clinical Practice
Brief Title: Study To Optimize Photodynamic Transurethral Resection of the Bladder (TUR-B) In Clinical Practice
Acronym: OPTIC-III
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: A-94-58150-002
Record Dates: First submitted 2013-11-28; First posted 2013-12-16 (Estimated); Last update posted 2019-08-16 (Actual); Status verified 2019-08

CONDITIONS: Photodynamic Transurethral Resection of the Bladder (TUR-B)
MeSH Terms: interventions — 5-aminolevulinic acid hexyl ester

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- TUR-B: TUR-B in patients suspected to have non-muscle-invasive bladder cancer (NMIBC).
  Interventions: Drug: Hexvix

INTERVENTIONS:
Drug: Hexvix — As this is a non-interventional study, detection of NMIBC with Hexvix is in a pre-defined group, chosen prior to and independently from the decision to enrol the subject in this study.
  The detection with Hexvix should be in accordance with local Summary of Product Characteristics [SmPC].
  Subjects will be treated in accordance with usual medical practice during their participation in this study, no additional assessment or tests will be required.
  Other Names: hexyl aminolevulinate (HAL)

SUMMARY:
The purpose of the study is to assess additional detection of Non-Muscle-Invasive Bladder Cancer (NMIBC) with hexyl aminolevulinate (HAL) cystoscopy based on lesions in patients undergoing TUR-B compared to white-light cystoscopy under the conditions of daily clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Indication of TURB due to suspicion of NMIBC (patients suspected to have non muscle invasive bladder cancer).
* Subject able to comply with the protocol.
* Written informed consent available.

Exclusion Criteria:

* Hypersensitivity to the active substance or to any of the excipients of the solvent.
* Porphyria.
* Gross haematuria.
* Women of child-bearing potential.
* Repeated TURB (control TURB) as part of follow-up after previous TURB.
* Bacillus Calmette-Guerin (BCG) or Mitomycin / intravesical chemotherapy instillation therapy in the last 12 weeks or any other contraindications according to the SmPC.
* Subjects not able to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Bladder cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2013-07; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Detection rate | At TUR-B visit, up to 1 year
  Detection rate is defined as number of lesions detected or not (Detection by HAL cystoscopy compared to white light cystoscopy confirmed by histology).

SECONDARY OUTCOMES:
Detection rate for risk groups according to the European Organisation for Research and Treatment of Cancer (EORTC)-score | At TUR-B visit, up to 1 year
  Risk groups are low, intermediate and high.
Evaluation of the diagnostic procedure in practice and compared to procedures according to published recommendations | At TUR-B visit, up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (2):
- Germany (2):
  - Caritas-Krankenhaus St. Josef, Klinik fuer Urologie, Regensburg
  - Klinikverbund Südwest, Sindelfingen